CLINICAL TRIAL: NCT06558747
Title: Comparison of the Clinical Success of Pediatric Zirconia Crowns Applied with Different Luting Cements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hüseyin Karayılmaz, Proffessor at Pediatric Dentistry, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDK-2016-1761
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries; Dental Plaque; Dental Caries in Children
MeSH Terms: conditions — Dental Caries; Dental Plaque | interventions — Cementation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Device: Bioactive Cement (Experimental): BioCem™ (NuSmile, Texas, USA) was evenly distributed to the inner surface of the crown with the syringe and immediately placed onto the teeth. Crowns were stabilized for 20 seconds before applying halogen/LED light (800-1200mW/cm2) (Valo Cordless, Ultradent) to the buccal and lingual/palatal surfaces for three seconds each.
  Interventions: Procedure: Tooth Preperation; Procedure: Cementation
- Device: Resin Cement (Experimental): The inner surface of the crowns was treated with 'G-Multi Primer' using a brush and subsequently air-dried. The surfaces of the prepared teeth were treated with 37% orthophosphoric acid. The tooth surfaces were rinsed with an air-water spray to remove the acid from the surfaces. After the etching process, the 'G-Premio Bond' was applied to the teeth surfaces with a brush, rubbed for 10 seconds, and then air-dried for five seconds. Then the teeth were exposed to halogen/LED light (800-1200mW/cm2) (Valo Cordless, Ultradent) for 10 seconds. G-CEM Linkforce (GC, USA) resin cement was gently applied to crowns, and then crowns were pressed onto the prepared teeth with finger pressure.
  Interventions: Procedure: Tooth Preperation; Procedure: Cementation
- Device: Glass-ionomer cement (Experimental): The capsule was attached to the mixer and mixed for 10 seconds. The cement was evenly distributed to the crowns paying attention that there were no air voids. Then crowns were placed by pressing them onto the prepared teeth with finger pressure.
  Interventions: Procedure: Tooth Preperation; Procedure: Cementation
- Device: Resin-modified glass-ionomer cement (Experimental): The cement was placed into the crown with the self-mixing syringe, ensuring no air voids were created. The crowns were then seated onto the teeth with finger pressure.
  Interventions: Procedure: Tooth Preperation; Procedure: Cementation

INTERVENTIONS:
Procedure: Tooth Preperation — After the caries were removed, the teeth were prepared by shaving according to the manufacturer's recommendations for NuSmile ZR.
Procedure: Cementation — Pediatric zirconia crowns were placed on the prepared teeth with finger pressure, following the manufacturer's instructions for the luting cement to be used. For each cement, the recommended setting time was observed, and excess cement residues were removed accordingly.

SUMMARY:
This randomized controlled trial aims to evaluate and compare the clinical outcomes of prefabricated zirconia crowns (PZCs) for primary molars cemented with different luting cements. The main questions to answer are:

Will there be any difference in the clinical success regarding retention among the PZCs cemented with different luting cements? Will there be any difference in the clinical success regarding periodontal health among the PZCs cemented with different luting cements? Will there be any difference in the clinical success regarding pulpal survival among the PZCs cemented with different luting cements? Fifty-three children (60 teeth), between 5 and 11 years old enrolled for the study. Researchers will compare the retention status, plaque index (PI), gingival index (GI), and probing depth (PD) scores, and endodontic/periodontal pathology of PZCs.

Participants will:

- visit the clinic 1st,3rd,6th,12th months after the restoration.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* no history of allergies
* a Frankl scale score of 3 or 4
* has at least one carious primary molar

Teeth:

* No percussion or palpation sensitivity
* No pathological root resorption
* No abscess and/or fistula
* No radiolucency at the furcation area
* No prior pulpal treatment
* Presence of permanent successor
* No mobility or periodontal disease
* Normal position of permanent successor
* An interproximal decay and/or extensive decay with at least 2 surfaces
* If present, physiological root resorption no more than one-third of the root
* Opposing teeth in occlusal contact
* Normal lamina dura and periodontal space

Exclusion Criteria:

* congenital and/or developmental defects
* history of bruxism
* skeletal and/or dental malocclusion
* history of trauma
* infraocclusion

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Retention Status | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  The clinical success of the crowns regarding the retention status was evaluated as either present or absent based on whether the crown remained on the restored tooth at each follow-up appointment. Crowns that were still in place during the follow-up visit were considered successful in terms of retention, while those that had decemented were considered unsuccessful.

SECONDARY OUTCOMES:
Pulpal Survival | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  Maintaining pulpal vitality is also a criterion for the success of a restoration and is assessed not by a graded score but by the presence or absence of symptoms and findings. In this study, pulpal vitality was clinically evaluated based on the presence or absence of percussion sensitivity, palpation sensitivity, gingival redness, fistula or abscess. If percussion sensitivity, palpation sensitivity, or the formation of a fistula or abscess were present, the restoration was classified as unsuccessful regarding pulpal vitality. In cases of gingival redness or unclear clinical symptoms, a periapical radiograph was taken. If presence or absence of radiolucency in the periapical or furcal area was detected in the radiograph, the restoration was classified as unsuccessful regarding pulpal vitality.
Plaque Index | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  The clinical success of a full-coverage restoration is also related to periodontal health. The impact of the luting cement on periodontal health was investigated by recording the plaque index (PI), at all follow-up visits. The PI was recorded based on the criteria established by Silness and Löe, with 0 being the best and 3 being the worst. The recorded scores were compared among the groups.
Gingival Index | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  The clinical success of a full-coverage restoration is also related to periodontal health. The impact of the luting cement on periodontal health was investigated by recording the gingival index (GI) at all follow-up visits. The GI were recorded based on the criteria established by Silness and Löe, with 0 being the best and 3 being the worst. The recorded scores were compared among the groups.
Probing Depth | Evaluations were conducted at the 1st, 3rd, 6th, 12th months.
  The clinical success of a full-coverage restoration is also related to periodontal health. The impact of the luting cement on periodontal health was investigated by measuring the probing depth (PD) of each crown at all follow-up visits. PD was measured using a universal periodontal probe by probing the gingival sulcus. The gingival sulcus is the space between the free gingiva and the tooth. It has a V-shape and allows the periodontal probe to enter. Clinically, a healthy gingival sulcus depth ranges from 0.5 to 2 mm on the buccal and lingual surfaces, while a pocket depth of up to 3 mm is considered normal in the proximal areas. A deeper pocket depth is considered an indication of periodontal disease. The recorded scores were compared among the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Dentistry, Akdeniz University, Antalya, Turkey (Türkiye)